CLINICAL TRIAL: NCT03487042
Title: Bimatoprost 0.03% Solution, NB-UVB and Fractional Carbon Dioxide Laser in Treatment of Generalized Vitiligo
Brief Title: Bimatoprost 0.03% Solution With NB-UVB Versus Their Use With Fractional Carbon Dioxide Laser in Treatment of Generalized Vitiligo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Hassan Ali, Principle investigator, Assiut University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BSNUFCO2
Record Dates: First submitted 2018-03-11; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Generalized Vitiligo
MeSH Terms: interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Generalized vitiligo patients (Experimental): Each patient with generalized vitiligo will be subjected to the following:
  One side will be treated by narrow band ultraviolet rays sessions twice weekly for 3 months + topical bimatoprost 0.03% ophthalmic solution solution twice daily ( 1 drop for each 2 cm2 ) and the other side will be treated by topical bimatoprost 0.03% ophthalmic solution twice daily ( 1 drop for each 2 cm2 ) + narrow band ultraviolet rays sessions twice weekly for 3 months + 10.600-nm fractional carbon dioxide laser sessions twice monthly for 3 months.
  Interventions: Drug: Bimatoprost 0.03% ophthalmic solution

INTERVENTIONS:
Drug: Bimatoprost 0.03% ophthalmic solution — Each patient will be subjected to the following:
  One side will be treated by narrow band ultraviolet rays B sessions twice weekly for 3 months + topical bimatoprost 0.03% solution twice daily ( 1 drop for each 2 cm2 ) and the other side will be treated by topical bimatoprost 0.03% twice daily ( 1 drop for each 2 cm2 ) + narrow band ultraviolet rays B sessions twice weekly for 3 months + 10.600-nm fractional carbon dioxide laser sessions twice monthly for 3 months.
  Patients' Evaluation:
  The recruited patients will be subjected to:
  A) Full history taking. B) General clinical examination. C) Dermatological examination of the skin lesions. D) Vitiligo area scoring index score will be calculated for each patient E) Clinical photographs will be taken at baseline, after each month during treatment and after the end of treatment by 3 months.
  F) A skin biopsy from the treated lesions for histochemical examination. F) Dermoscopic evaluation of the treated sites every 2 weeks.
  Other Names: Narrow band ultraviolet rays B; Fractional carbon dioxide laser

SUMMARY:
Vitiligo is a chronic disorder of pigmentation characterized by the development of white macules on the skin due to loss of epidermal melanocytes. It affects approximately 0.5%-2% of general population world-wide, without predilection for sex or race.Vitiligo can be classified into segmental or non-segmental. Non-segmental or generalized vitiligo is the most common clinical presentation and often involves the face and acral regions.

Multiple monotherapy modalities are established to treat vitiligo but the response is variable, unsatisfactory, and requiring a prolonged course. This problem is exaggerated by the multifactorial and polygenic nature of the pathomechanism of the disease. These facts pave the way to combination therapy that showed better and safe repigmentation response than monotherapy.

DETAILED DESCRIPTION:
Bimatoprost 0.03% ophthalmic solution is a synthetic prostaglandin F2 alpha analog that is approved for the treatment of glaucoma and eyelashes hypotrichosis (Lee et al, 2017). Cutaneous hyperpigmentation of the treated sites has been reported as a side effect with this agent. Phototherapy (narrow band ultraviolet B (NB-UVB)) of wavelength 308 nm, is considered as a successful method of treatment of vitiligo. The cytotoxic T-cells accountable for the destruction of melanocytes and disappearance of melanin are eliminated by phototherapy through apoptosis (diffuse repigmentation) and UVB does stimulate melanocytic proliferation and their migration to the epidermis from nearby follicular units (follicular repigmentation) and perilesional active melanocytes (marginal repigmentation).

In recent years, fractional carbon dioxide laser has been introduced as an add-on treatment for vitiligo. It represents a new modality for skin resurfacing based on the theory of fractional photothermolysis. The beneficial effect of fractional carbon dioxide laser on vitiligo is the release of cytokines and growth factors that act as mitogens for melanogenesis. It also alters the skin barrier, which results in increased penetration of topical drugs and ultraviolet (UV) radiation, so it can be used in combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 12.
2. Patients with non-segmental vitiligo.
3. Lesions stable for at least one year.
4. Patients who were unresponsive to medical treatment or photo therapy for at least 3 months.
5. No sex or site predilection.
6. Bilateral and symmetrical lesions with maximum size of 10×10 cm.

Exclusion Criteria:

1. Patients with active infection.
2. Patients with sensitivity to bimatoprost or photosensitivity.
3. Patients with history or active skin cancer.
4. Pregnant or lactating females.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Repigmentation of skin lesions | 3 months
  Patients will be followed up by two blind dermatologists after 3 months to detect:
  The percent of repigmentation: that will be subjectively rated with a previously reported scoring system:
  * < 25% repigmentation (poor).
  * 25-50% repigmentation (fair).
  * 50-75% repigmentation (good). -> 75% repigmentation (excellent).
Frequency and types of side effects | 3 months
  Frequency and types of side effects.

SECONDARY OUTCOMES:
Vitiligo area scoring index score | 3 months
  Vitiligo area scoring index score percent change will be calculated by subtracting the pre- procedure vitiligo area scoring index score from the post-procedure vitiligo area scoring index score and dividing by the pre-procedure vitiligo area scoring index score.
Patient satisfaction | 6 months
  The patient overall satisfaction will be assessed after 6 months according to Wong Overall satisfaction:
  1. dissatisfied
  2. neutral
  3. somewhat satisfied
  4. moderately satisfied
  5. very satisfied

REFERENCES:
- [Background] Ezzedine K, Eleftheriadou V, Whitton M, van Geel N. Vitiligo. Lancet. 2015 Jul 4;386(9988):74-84. doi: 10.1016/S0140-6736(14)60763-7. Epub 2015 Jan 15. PMID 25596811
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315
- [Background] Abdelghani R, Ahmed NA, Darwish HM. Combined treatment with fractional carbon dioxide laser, autologous platelet-rich plasma, and narrow band ultraviolet B for vitiligo in different body sites: A prospective, randomized comparative trial. J Cosmet Dermatol. 2018 Jun;17(3):365-372. doi: 10.1111/jocd.12397. Epub 2017 Aug 20. PMID 28834191
- [Background] Lee D, Mantravadi AV, Myers JS. Patient considerations in ocular hypertension: role of bimatoprost ophthalmic solution. Clin Ophthalmol. 2017 Jul 10;11:1273-1280. doi: 10.2147/OPTH.S118689. eCollection 2017. PMID 28744094
- [Background] Bagherani N, Smoller BR. Efficacy of bimatoprost in the treatment of non-facial vitiligo. Dermatol Ther. 2017 Mar;30(2). doi: 10.1111/dth.12409. Epub 2016 Aug 23. No abstract available. PMID 27550870
- [Background] Salah Eldin MM, Sami NA, Aly DG, Hanafy NS. Comparison Between (311-312 nm) Narrow Band Ultraviolet-B Phototherapy and (308 nm) Monochromatic Excimer Light Phototherapy in Treatment of Vitiligo: A Histopathological Study. J Lasers Med Sci. 2017 Summer;8(3):123-127. doi: 10.15171/jlms.2017.22. Epub 2017 Jun 27. PMID 29123631
- [Background] Omi T, Numano K. The Role of the CO2 Laser and Fractional CO2 Laser in Dermatology. Laser Ther. 2014 Mar 27;23(1):49-60. doi: 10.5978/islsm.14-RE-01. PMID 24771971
- [Background] Kim HJ, Hong ES, Cho SH, Lee JD, Kim HS. Fractional Carbon Dioxide Laser as an "Add-on" Treatment for Vitiligo: A Meta-analysis with Systematic Review. Acta Derm Venereol. 2018 Feb 7;98(2):180-184. doi: 10.2340/00015555-2836. PMID 29110015
- [Background] Wong L, Vasconez HC. Patient satisfaction after Nd:YAG laser-assisted lipolysis. Ann Plast Surg. 2011 May;66(5):561-3. doi: 10.1097/SAP.0b013e31820b3d1e. PMID 21451378